CLINICAL TRIAL: NCT06260397
Title: Ultrasound Guided Serratus Anterior Plane Block Versus Costotransverse Block on Postoperative Analgesia and Safety Following Modified Radical Mastectomy Surgeries
Brief Title: Serratus Anterior Plane Block and Costotransverse Block for Analgesia Following Modified Radical Mastectomy Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: analgesia for MRM surgeries
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-01

CONDITIONS: Regional Anesthesia Morbidity
MeSH Terms: interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- serratus anterior plane block (Experimental): while the patients in lateral position, serratus anterior plane block will be done using high frequency linear ultrasound probe at the level of fourth rib.30 ml of 0.25% bupivacaine will be injected.
  Interventions: Procedure: serratus anterior plane block
- costotransverse plane block (Experimental): while the patients in lateral position, costotransverse block will be done using 22-gauge echogenic needle. the needle is advanced in-plane lateral to the spinous process of the 4th thoracic vertebra from caudally cephalad.30 ml of 0.25% bupivacaine will be injected
  Interventions: Procedure: costotransverse block
- patient controlled analgesia (Experimental): After successful extubation, patients will be transferred to PACU. Patients will receive a bolus dose of 5 mg nalbuphine then PCA pump in the form of 20 mg nalbuphine HCL in 100 ml 0.9% normal saline with basal rate of infusion 5ml/hr with self-administration bolus of 0.5ml with 15 min lock-out time.
  Interventions: Procedure: patient controlled analgesia

INTERVENTIONS:
Procedure: serratus anterior plane block — using ultrasound, 30 ml of bupivacaine 0.25% will be injected in the plane between the latissimus dorsi and serratus muscles
  Arms: serratus anterior plane block
Procedure: costotransverse block — using ultrasound, 30 ml of bupivacaine 0.25% will be injected in the costotransverse plane of fourth rib
  Arms: costotransverse plane block
Procedure: patient controlled analgesia — PCA pump in the form of 20 mg nalbuphine HCL in 100 ml 0.9% normal saline with basal rate of infusion 5ml/hr. with self-administration bolus of 0.5ml with 15 min lock-out time.
  Arms: patient controlled analgesia

SUMMARY:
Adequate pain management following modified radical mastectomy (MRM) is crucial for early ambulation and patient satisfaction. Breast cancer is the most common malignancy in females, with an increasing incidence in recent years. Surgery is one of the mainstays of therapy for breast cancer, and modified radical mastectomy (MRM) is the most effective and common type of invasive surgical treatment. Post-mastectomy pain syndrome (PMPS) is a surgical complication of breast surgery characterized by chronic neuropathic pain. The aim of this study is to investigate the efficacy and safety of single injection CTB versus SAPB on post-operative acute pain as a part of a multimodal analgesia plan in patients undergoing MRM.

DETAILED DESCRIPTION:
Patients will be divided randomly by the computer into three groups, group (A): will receive serratus anterior plane block, group (B): will receive costotransverse block and group(C): patient controlled analgesia group (PCA).

Group (A) (SAPB):

SAPB will be performed using an ultrasound machine with a high-frequency linear probe . All patients will be in lateral position to perform the block. At the level of the fourth rib with 45-degree angle, targeting the plane between the latissimus dorsi and serratus muscles, SAPB block will be performed unilaterally on the ipsilateral side of surgery.

Group (B) (CTB):

CTB will be performed using an ultrasound machine with a high-frequency linear probe. All patients will be in lateral position to perform the block. CTB block will be performed unilaterally on the ipsilateral side of surgery at the level of fourth rib.

Group (C) (patient controlled analgesia):

After successful extubation, patients will be transferred to PACU. Patients will receive a bolus dose of 5 mg nalbuphine then PCA pump in the form of 20 mg nalbuphine HCL in 100 ml 0.9% normal saline with basal rate of infusion 5ml/hr with self-administration bolus of 0.5ml with 15 min lock-out time.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anaesthesiologists (ASA) Physical Status Class I, II.
2. Scheduled for modified radical mastectomy (MRM).
3. Body weight ranging from 60 to 100 kilograms.

Exclusion Criteria:

1. Declining to give a written informed consent.
2. History of allergy to the medications used in the study.
3. Contraindications to regional anesthesia (including patient: refusal, coagulopathy, and local infection).
4. Psychiatric disorders.
5. Significant cognitive dysfunction.
6. American Society of Anesthesiologists (ASA) Physical Status Class III and IV.
7. Daily use of opioids.
8. Obesity (BMI > 35 kg/m2).

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2023-12-28 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale score at 0,6,12 and 24 hour post-operatively. visual analogue scale is a scale from 0 to 10, 0 represent no pain at all and 10 represent the worst pain | 24 hour post-operative
  Visual Analogue Scale score will be assessed at both rest and arm elevation

SECONDARY OUTCOMES:
The total dose of nalbuphine consumption is used postoperatively per patient rescue analgesia for 24. | 24 hour post-operative
  dose of nalbuphine consumed by patients
Incidence of chronic pain after 6 months of surgery | 6 months after surgery
  How many people develop chronic pain after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- AinShamsU, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao Y, Jin W, Pan P, Feng S, Fu D, Yao J. Ultrasound-guided transversus thoracic muscle plane-pectoral nerve block for postoperative analgesia after modified radical mastectomy: a comparison with the thoracic paravertebral nerve block. Perioper Med (Lond). 2022 Jul 27;11(1):39. doi: 10.1186/s13741-022-00270-3. PMID 35883207
- [Background] Aygun H, Kiziloglu I, Ozturk NK, Ocal H, Inal A, Kutlucan L, Gonullu E, Tulgar S. Use of ultrasound guided single shot costotransverse block (intertransverse process) in breast cancer surgery: a prospective, randomized, assessor blinded, controlled clinical trial. BMC Anesthesiol. 2022 Apr 18;22(1):110. doi: 10.1186/s12871-022-01651-3. PMID 35436844
- [Background] Holm UHU, Andersen CHS, Hansen CK, Tanggaard K, Borglum J, Nielsen MV. Ultrasound-guided multiple-injection costotransverse block for mastectomy and primary reconstructive surgery. A study protocol. Acta Anaesthesiol Scand. 2022 Mar;66(3):386-391. doi: 10.1111/aas.14018. Epub 2022 Jan 5. PMID 34907523
- [Background] Jack JM, McLellan E, Versyck B, Englesakis MF, Chin KJ. The role of serratus anterior plane and pectoral nerves blocks in cardiac surgery, thoracic surgery and trauma: a qualitative systematic review. Anaesthesia. 2020 Oct;75(10):1372-1385. doi: 10.1111/anae.15000. Epub 2020 Feb 16. PMID 32062870
- [Background] Sahin A, Baran O, Gultekin A, Yildirim I, Arar C, Gunkaya M. Serratus anterior plane block for tertiary revision rhinoplasty with rib cartilage harvest. J Clin Anesth. 2021 Oct;73:110292. doi: 10.1016/j.jclinane.2021.110292. Epub 2021 Apr 29. No abstract available. PMID 33934036
- [Background] Ohgoshi Y, Usui Y, Ando A, Takeda Y, Ohtsuka A. Injection at the costotransverse notch facilitates paravertebral spread of the erector spinae plane block: A cadaveric study. J Clin Anesth. 2020 May;61:109630. doi: 10.1016/j.jclinane.2019.109630. Epub 2019 Oct 23. No abstract available. PMID 31668466
- [Background] Wang Y, Shi M, Huang S, He X, Gu X, Ma Z. Ultrasound-guided serratus anterior plane block versus paravertebral block on postoperation analgesia and safety following the video-assisted thoracic surgery: A prospective, randomized, double-blinded non-inferiority clinical trial. Asian J Surg. 2023 Oct;46(10):4215-4221. doi: 10.1016/j.asjsur.2022.11.125. Epub 2022 Dec 12. PMID 36517403